CLINICAL TRIAL: NCT00004058
Title: Phase I Study of 12-O-tetradecanoylphorbol-13-acetate (TPA) in Patients With Refractory Hematologic Malignancies/Bone Marrow Disorders
Brief Title: 12-O-Tetradecanoylphorbol-13-acetate in Treating Patients With Hematologic Cancer or Bone Marrow Disorder
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: At this time it is felt that we will not gain further information from an additional patients.
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Roger Strair, MD, PhD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Purpose: Treatment
Other Study IDs: 5986; CDR0000067255; P30CA072720 (NIH); CINJ-059806; UMDNJ-2716; NCI-G99-1573
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Precancerous/Nonmalignant Condition
Keywords: monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; refractory hairy cell leukemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system lymphoma; prolymphocytic leukemia; primary systemic amyloidosis; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; refractory cytopenia with multilineage dysplasia; recurrent mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Tetradecanoylphorbol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tetradecanoylphorbol acetate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of 12-O-tetradecanoylphorbol-13-acetate in treating patients with hematologic cancer or bone marrow disorder that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose limiting toxicity of 12-O-tetradecanoylphorbol-13-acetate (TPA) in patients with relapsed or refractory hematologic malignancies or bone marrow disorders.
* Determine the pharmacokinetics of TPA in these patients.
* Determine the effects of TPA on the cellular composition of blood and bone marrow in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive 12-O-tetradecanoylphorbol-13-acetate (TPA) IV over 1 hour on days 1 and 8 followed by 2 weeks of rest. Courses repeat in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of TPA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven relapsed or refractory hematologic malignancy or bone marrow disorder for which there is no standard curative therapy, including, but not limited to:

  * Myelodysplasia
  * Multiple myeloma
  * Myeloproliferative syndrome
  * Chronic lymphocytic leukemia
  * Aplastic anemia
  * Non-Hodgkin's lymphoma
  * Acute leukemia
  * Hodgkin's lymphoma
  * Chronic myelogenous leukemia

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 1 month

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* Cardiac ejection fraction greater than 40%

Pulmonary:

* FEV_1 greater than 50% predicted

Other:

* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 10 weeks after study participation
* No uncontrolled psychiatric or medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Greater than 3 weeks since prior biologic therapy

Chemotherapy:

* Greater than 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States